CLINICAL TRIAL: NCT06498479
Title: ARTEMIS-008：A Multicenter, Randomized, Open-label, Phase 3 Study of HS-20093 Compared With Topotecan in Subjects With Relapsed Small Cell Lung Cancer After Platinum-based First-line Chemotherapy
Brief Title: ARTEMIS-008：HS-20093 Compared With Topotecan in Subjects With Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-301
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS-20093 (Experimental): Participants will receive HS-20093 as an intravenous (IV) infusion at dose of 8.0 mg/kg on Day 1 of each 21-day cycle until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: HS-20093
- Topotecan (Active Comparator): Participants will receive topotecan until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: HS-20093 — HS-20093 will be administered as an IV infusion at dose of 8.0 mg/kg on Day 1 of each 21-day cycle.
  Arms: HS-20093
Drug: Topotecan — Topotecan will be administered per drug label.
  Arms: Topotecan

SUMMARY:
The main objective of this study is to compare the efficacy of HS-20093 with standard of care (SOC) on prolonging overall survival (OS) in subjects with relapsed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
This is a phase 3, randomized, open-label, multicenter study comparing HS-20093 with topotecan in patients with limited or extensive SCLC that had disease progression on or after first-line platinum-based regimen. Subjects will be randomized by a ratio of 1:1 to receive HS-20093 or topotecan until disease progression.

The primary objective of this study is to assess whether treatment with HS-20093 prolongs OS compared with treatment of topotecan among subjects with relapsed SCLC.

The secondary objectives of the study are to further evaluate the efficacy/safety of HS-20093. The exploratory objectives are to characterize the pharmacokinetics of HS-20093, evaluate E-R relationship, immunogenicity of HS-20093, B7-H3 protein expression and soluble B7-H3 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age.
2. Histologically or cytologically confirmed SCLC.
3. Subjects who progressed on or after first-line platinum-based regimens.
4. Has at least 1 measurable lesion as defined per RECIST 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Minimum life expectancy of more than 12 weeks.
7. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential.
8. Men or women should be using adequate contraceptive measures throughout the study.
9. Subject has provided informed consent/assent prior to initiation of any study specific activities/procedures.

Exclusion Criteria:

1. Combined SCLC, any previous diagnosis of transformed SCLC or SCLC that has transformed to NSCLC.
2. Chemotherapy-free interval ≤30 days.
3. Has received prior treatment with anti-B7 homologue 3 (B7-H3) targeted agents.
4. Has received prior treatment with topoisomerase I inhibitor, including ADC that consists of topoisomerase I inhibitor.
5. Has inadequate washout period before randomization as specified in the protocol.
6. Untreated or symptomatic brain metastases with exceptions defined in the protocol.
7. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 with exceptions defined in the protocol.
8. History of other malignancy with exceptions defined in the protocol.
9. Inadequate bone marrow reserve or organ dysfunction.
10. Evidence of cardiovascular risks.
11. Severe, uncontrolled or active cardiovascular diseases.
12. Severe or uncontrolled diabetes.
13. Severe or uncontrolled high blood pressure.
14. Clinically significant bleeding or obvious bleeding tendency within 1 month before randomization.
15. Severe arterial or venous thromboembolic events within 3 months prior to randomization.
16. Severe infections within 4 weeks before randomization.
17. Receiving systemic corticosteroid therapy within 30 days prior to randomization with exceptions defined in the protocol.
18. The presence of active infectious diseases before randomization.
19. Current hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.
20. History of interstitial lung disease, immunotherapy-induced pneumonitis, clinically moderate or severe pulmonary disease.
21. History of severe neuropathy or mental disorders.
22. Female subjects of childbearing potential; female subjects who are breastfeeding or who plan to breastfeed while on study; female subjects planning to become pregnant while on study.
23. Vaccination or hypersensitivity of any level within 4 weeks before randomization.
24. History of severe hypersensitivity reaction, severe infusion reaction or allergy to recombinant human or mouse derived proteins.
25. Hypersensitivity to any ingredient of HS-20093, DNA topoisomerase I inhibitor or regimens of Topotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death due to any cause; Up to approximately 4.5 years
  Overall survival is defined as the time interval from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Assessed by Blinded Independent Central Review and Investigators | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 4.5 years.
  Confirmed ORR is defined as the sum of the complete response (CR) rate and partial response (PR) rate as per BICR and investigator per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Disease Control Rate (DCR) Assessed by Blinded Independent Central Review and Investigator | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 4.5 years.
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) per BICR and investigator assessment per RECIST v1.1.
Duration of Response Assessed by Blinded Independent Central Review and Investigator | From the date of first documentation of confirmed response (CR or PR) to the first documentation of objective progression or to death due to any cause, whichever occurs first; Up to approximately 4.5 years.
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death.
Progression-free Survival Assessed by Blinded Independent Central Review and Investigator | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 4.5 years.
  PFS is defined as the time interval from the randomization to disease progression as per BICR and investigator assessment or death due to any cause.
Incidence and Grade of Participants With Treatment-emergent Adverse Events | From the date of first dose to the end of safety follow-up; Up to approximately 4.5 years.
  TEAEs are assessed based on NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliate Hospital of GUANGZHOU Medical University, Guangzhou
  - Tongji Hospital, Wuhan